CLINICAL TRIAL: NCT05566561
Title: Postoperative Analgesic Efficacy of Ultrasound-guided Para-sartorial Compartment Block in Knee Surgery: A Randomized Study
Brief Title: Para-sartorial Compartment Block in Knee Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Primary researcher, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 31
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis; Knee Injuries; Knee Disease; Knee Arthritis
Keywords: Knee Surgery; Postoperative pain management; Postoperative Analgesia; Parasartorial compartment block
MeSH Terms: conditions — Osteoarthritis, Knee; Knee Injuries

STUDY DESIGN:
Intervention Model Description: There are two models for this study. Parasartorial compartment block (PSCB) group, and control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the outcomes assessor who performs postoperative pain evaluation will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group PSCB = Parasartorial compartment block group (Active Comparator): After placing the linear ultrasound probe in the middle of the anterior superior line to the patella and spina drug, the probe will be advanced cephalad to visualize the intermediate femoral cutaneous nerve over the satrorious. Then the block will be applied. Three injections will be made with a single needle entry in the same imaging. The procedure will be completed by applying the first injection to the femoral triangle (10 ml of local anesthetic solution), the second injection to the subsartorial region (10 ml of local anesthetic solution) lateral to the femoral artery, and the third injection to the suprasartorial region (10 ml of local anesthetic solution) (total 30 ml of 0.25% solution). concentration bupivacaine). The block location will be confirmed by injecting 2 ml of saline in every three injections.
  Interventions: Drug: Postoperative analgesia management
- Group C = Control group (Active Comparator): Wound infiltration will be applied by the surgical team
  Interventions: Drug: Postoperative analgesia management

INTERVENTIONS:
Drug: Postoperative analgesia management — Intravenous 0.5 mg/kg tramadol and 400 mg ibuprofen will be administered to all patients 30 minutes before the end of the surgical procedure. In the postoperative period, patients will be administered ibuprofen iv 400 mg 3x1. Postoperative patient evaluation will be performed by another pain nurse who is unaware of the procedure. Patients in all groups will be attached to IV PCA containing 10 mcg/ml fentanyl, 10 mcg bolus without infusion dose, and 10 min lock time protocol. If the NRS score is ≥ 4, 0.5 mg kg-1 iv meperidine will be administered as a rescue analgesic.

SUMMARY:
Selective blockade of the saphenous nerve branches is among the regional anesthesia techniques in knee surgery. In this block, analgesia is provided without motor block and is an essential advantage in terms of early mobilization in the postoperative period. Blockage of motor branches causes a delay in mobilization and increases the risk of falling. The vastus medialis and its medical femoral cutaneous branch are rich in the femoral triangle. Effective postoperative analgesia is provided by a femoral triangle (triangle) blockade. The intermediate femoral cutaneous nerve courses over the sartorius muscle. Anatomically, the femoral triangle follows a separate path. When the femoral triangle and the blockade of the intermediate femoral cutaneous nerve are combined, it is called PSKB block. Parasartorial compartment block (PSKB); is based on the blockade of the branches of the saphenous nerve, the two largest sensory nerves from the femoral nerve to the knee, and is predicted to provide effective postoperative analgesia in knee arthroplasty.

DETAILED DESCRIPTION:
Selective blockade of the saphenous nerve branches is among the regional anesthesia techniques in knee surgery. In this block, analgesia is provided without motor block and is an essential advantage in terms of early mobilization in the postoperative period. Blockage of motor branches causes a delay in mobilization and increases the risk of falling. The vastus medialis and its medical femoral cutaneous branch are rich in the femoral triangle. Effective postoperative analgesia is provided by a femoral triangle (triangle) blockade. The intermediate femoral cutaneous nerve courses over the sartorius muscle. Anatomically, the femoral triangle follows a separate path. When the femoral triangle and the blockade of the intermediate femoral cutaneous nerve are combined, it is called PSKB block. Parasartorial compartment block (PSKB); is based on the blockade of the branches of the saphenous nerve, the two largest sensory nerves from the femoral nerve to the knee, and is predicted to provide adequate postoperative analgesia in knee arthroplasty.

Pascarella et al. applied PSKB to a 58-year-old patient who underwent knee surgery under spinal anesthesia and had pain in the postoperative period and reported that the patient with a visual pain score of 9 decreased to 2 after the block.

This study, it is aimed to evaluate the effectiveness of para-sartorial canal block for postoperative analgesia management in patients undergoing knee surgery. Our primary aim is to compare postoperative opioid consumption, and our secondary aim is to evaluate postoperative pain scores (Numerical rating scale-NRS), the presence of motor blockade, first postoperative mobilization time, and side effects (allergic reaction, nausea, vomiting, etc.) associated with opioid use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA classification I-III,
* Aged 18-75 years
* Who will be scheduled for knee surgery under spinal anesthesia.

Exclusion Criteria:

* Patients who have a history of bleeding diathesis,
* Take anticoagulant therapy,
* History of chronic pain before surgery,
* Multiple trauma,
* Who cannot assess their pain,
* Who have been operated under spinal anesthesia,
* Who have an infection in the area and do not accept the procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2025-08-10 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Pain scores (Numerical Rating Scale-NRS) | Changes from baseline pain scores at postoperative 8th hour
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)

SECONDARY OUTCOMES:
Rescue analgesia (Opioid-tramadol consumption) | Changes from baseline opioid consumption at postoperative 1, 2, 4, 8, 16 and 24 hours.
  The tramadol consumption as rescue analgesia will be evaluated
Adverse events will be recorded | Postoperative 24 hours period
  Adverse events; nausea, vomiting, itching

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators will not share IPD

REFERENCES:
- [Background] Pascarella G, Costa F, Del Buono R, Strumia A, Cataldo R, Agro F, Carassiti M. The para-sartorial compartments (PASC) block: a new approach to the femoral triangle block for complete analgesia of the anterior knee. Anaesth Rep. 2022 May 5;10(1):e12165. doi: 10.1002/anr3.12165. eCollection 2022 Jan-Jun. No abstract available. PMID 35547556
- [Background] Martin R, Kirkham KR, Ngo THN, Gonvers E, Lambert J, Albrecht E. Combination of femoral triangle block and infiltration between the popliteal artery and the capsule of the posterior knee (iPACK) versus local infiltration analgesia for analgesia after anterior cruciate ligament reconstruction: a randomized controlled triple-blinded trial. Reg Anesth Pain Med. 2021 Sep;46(9):763-768. doi: 10.1136/rapm-2021-102631. Epub 2021 May 26. PMID 34039734
- [Background] Stebler K, Martin R, Kirkham KR, Lambert J, De Sede A, Albrecht E. Adductor canal block versus local infiltration analgesia for postoperative pain after anterior cruciate ligament reconstruction: a single centre randomised controlled triple-blinded trial. Br J Anaesth. 2019 Aug;123(2):e343-e349. doi: 10.1016/j.bja.2019.04.053. Epub 2019 May 24. PMID 31130273